CLINICAL TRIAL: NCT07057674
Title: A Bioequivalence Study of HS-20094 Multi-dose Pre-filled Injection and HS-20094 Single-dose Pre-filled Injection in Overweight or Obese Participants
Brief Title: A Study of HS-20094 in Overweight or Obese Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HS-20094-106
Record Dates: First submitted 2025-06-02; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T1 group (Experimental): HS-20094 AI pen administered subcutaneously (SC) once a week.
  Interventions: Drug: HS-20094 AI pen;
- T2 group (Experimental): HS-20094 MDV pen administered subcutaneously (SC) once a week.
  Interventions: Drug: HS-20094 MDV pen

INTERVENTIONS:
Drug: HS-20094 AI pen; — Arm 1: Administered SC The dose is escalated every 4 weeks until the target dose of 15 mg is reached. The dose escalation scheme is as follows: 2.5 mg → 5 mg → 7.5 mg → 10 mg → 12.5 mg → 15 mg.
  Arms: T1 group
Drug: HS-20094 MDV pen — The dose is escalated every 4 weeks until the target dose of 15 mg is reached. The dose escalation scheme is as follows: 2.5 mg → 5 mg → 7.5 mg → 10 mg → 12.5 mg → 15 mg.
  Arms: T2 group

SUMMARY:
This is a multicenter, randomized, open-label, parallel clinical study to evaluate the bioequivalence of the HS-20094 MDV pen and AI pen in overweight or obese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the procedures and methods of this study, willing to strictly adhere to the clinical study protocol to complete this study, and voluntarily sign the informed consent form;
2. Adult male or female participants (aged 18-65 years (inclusive), calculated based on the date of signing the informed consent form);
3. Body mass index (BMI) ≥24.0 kg/m2 (BMI = weight (kg) / height2 (m2)); body weigh ≥45 kg for female participants and ≥50 kg for male participants.
4. Self-reported diet/exercise control alone for at least 12 weeks prior to screening, with a weight change of ≤5% in the past 12 weeks (based on self-report); calculation formula for weight change: (highest weight - lowest weight within 12 weeks prior to screening) ∕ highest weight * 100%;
5. Agree to take effective contraceptive measures from the signing of the informed consent form until 8 weeks after the last dose, and have no plans for conception or sperm/egg donation during this period (only non-drug contraceptive measures are permitted during the study).

Exclusion Criteria:

Participants with any of the following examination abnormalities at screening:

1. Laboratory test results meet any of the following criteria (if there is a clear reason for retesting, one re-examination can be conducted within the time window of the screening period, and the results of this re-examination will be used as the basis for screening):

   * HemoglobinA1c (HbA1c) ≥6.5% or fasting plasma glucose ≥7.0 mmol/L;

     * Fasting plasma glucose <2.8 mmol/L;

       * Alanine aminotransferase > 3 × ULN, or aspartate aminotransferase > 3 × ULN, or total bilirubin > 1.5 × ULN;

         * Triglyceride >500 mg/dL (5.64 mmol/L);

           * Estimated glomerular filtration rate (absolute eGFR) based on the CKD-EPI equation <60 mL/min;

             * Serum calcitonin level ≥50 ng/L; ⑦ Thyroid-stimulating hormone >6.0 mIU/L or <0.4 mIU/L;

               ⑧ Blood amylase or blood lipase >2×ULN;
               * Prothrombin time (PT)-international normalized ratio (INR) exceeds the upper limit of normal, and the investigator determines the abnormality to be clinically significant, making it unsuitable for the participant to be enrolled; ⑩ Hemoglobin <110 g/L (male) or <100 g/L (female); ⑪ Positive test result for any one or more of the following items: hepatitis B surface antigen, hepatitis C antibody, HIV antibody/p24 antigen, or Treponema pallidum antibody;

   Presence of any of the following diseases or medical history prior to screening or randomization:
2. Participants who currently have or with history of severe diseases involving nervous system, psychiatric system, digestive system, circulatory system, respiratory system, urinary system, etc., or have newly developed diseases before administration of the investigational product, and therefore are deemed by the investigator as unsuitable for participation in this study;
3. Past history or ultrasound findings during screening period include any of the following conditions: medical history of chronic pancreatitis, acute pancreatitis, cholecystitis, or symptomatic/treatment-requiring gallbladder stones (except for participants who have undergone cholecystectomy but are deemed eligible for enrollment by the investigator);
4. Participants with a history or family history of thyroid C-cell tumors or multiple endocrine neoplasia type 2;
5. Participants with a history of metabolic disorders (such as unexplained recurrent hypoglycemia) who are deemed unsuitable for participation in this study upon the evaluation by the investigator;
6. Presence of endocrine diseases or medical history that may significantly affect weight (e.g., Cushing's syndrome, hypothyroidism, hyperthyroidism, etc., except for hypothyroidism if thyroid hormone replacement dosage has been stabilized for at least 6 months), or obesity due to a single gene mutation or hereditary obesity syndrome, etc.;
7. Presence of autoimmune disorders and planned use of systemic glucocorticoid therapy or immunosuppressive therapy during the study;
8. Participants with a history of significant gastric emptying abnormalities, severe gastrointestinal disorder, or gastrointestinal surgery (excluding polypectomy, appendicectomy, and haemorrhoid operation) who are deemed unsuitable for participation in this study upon the evaluation by the investigator;
9. Participants who have undergone surgeries that may affect drug absorption, distribution, metabolism, or excretion, and are deemed unsuitable for enrollment by the investigator;
10. Participants who are prone to allergic reactions or with allergic constitution (e.g., those allergic to pollen, two or more drugs/foods), or participants with known hypersensitivity to any component of the investigational product or similar drugs (Tirzepatide, GLP-1R agonists, or compounds containing GLP-1R agonists); or participants with a history of photosensitivity.
11. Blood donation and/or blood loss ≥400 mL or bone marrow donation within 3 months prior to screening; or haemoglobinopathy, haemolytic anaemia, or sickle cell anaemia at screening;
12. Past medical history of moderate to severe depression; or history of suicidal ideation or suicidal behavior; or past medical history of serious psychiatric disorders, e.g., schizophrenia, bipolar affective disorder, etc.; or a score of ≥9 on the Patient Health Questionnaire-9 (PHQ-9) at screening (self-rated by the participant);

    Participants who received any of the following drugs or treatments prior to screening:
13. Participants who have been previously treated with similar drugs of HS-20094 (Tirzepatide, GLP-1 analogues, or related compounds), and/or those who require the use of DPP-4 inhibitors (drugs affecting GLP-1 levels) during the study;
14. Any use of drugs or treatments that may cause significant weight gain or loss within 3 months prior to screening:

    ① Use of any GLP-1R-related single/multi-target drug that promotes weight loss, including, but not limited to, GLP-1R agonists, glucagon-like peptide-1 receptor/glucagon receptor (GLP-1R/GCGR) agonists, glucagon-like peptide-1 receptor/glucose-dependent insulinotropic polypeptide receptor (GLP-1R/GIPR) agonists, GLP-1R/GIPR/GCGR agonists, etc.;

    ② Any drug that may cause weight gain, including: systemic glucocorticoid medications (except for short-term use of <14 days or topical administration, inhalation, intraocular, or nasal administration), tricyclic antidepressants, atypical antipsychotics, and mood stabilizers (e.g., imipramine, amitriptyline, mirtazapine, paroxetine, phenelzine, chlorpromazine, thioridazine, clozapine, olanzapine, valproate, valproate derivatives, lithium salts), etc.;

    ③ Any Chinese herbal medicines, health care products, meal replacements, weight-reducing teas, etc. or similar products for the purpose of weight loss;

    ④ Any approved or unapproved weight-reducing drugs, such as sibutramine hydrochloride, orlistat, phentermine, phenylpropanolamine, mazindol, phentermine, diethylpropion, lorcaserin, phentermine/topiramate coformulation, naltrexone/bupropion coformulation, etc.;

    ⑤ Any glucose-lowering drugs, such as metformin, sodium-glucose cotransporter-2 (SGLT2) inhibitors, thiazolidinediones (TZDs), etc.;
15. History of bariatric/metabolic surgery within 12 months prior to screening, or participants who have not recovered from any surgery or trauma at screening, or participants who have recovered from gastrointestinal surgery prior to screening that affected gastrointestinal motility;
16. Participants who have received immunization of any vaccine within four weeks prior to the first dose of the investigational product, or who plan to receive immunization of any vaccine during the study or within 2 weeks after study completion.
17. Participants who have participated in any other clinical studies and received administration of investigational products within 3 months prior to screening; or the time interval from administration in the previous clinical study is less than 7 half-lives (whichever is longer);

    Participants with any of the following conditions:
18. Participants with abnormal findings in physical examination, vital signs, clinical laboratory tests, abdominal ultrasound, thyroid color Doppler ultrasound, etc., deemed by the investigator to be clinically significant and assessed as unsuitable for enrollment.
19. Participants with heart rate (HR) of <50 beats per minute or >100 beats per minute by 12-lead electrocardiogram (ECG) during screening. A retest is allowed, and the participant will be excluded if both tests fail;
20. Presence of any of the following abnormalities on 12-lead ECG at screening: second or third degree AV block, long QT syndrome, pre-excitation syndrome, ventricular tachycardia, atrial fibrillation, or QTcF >450 ms in males and >470 ms in females, or any other arrhythmia deemed clinically significant by the investigator. Participants with abnormal QTcF on the first examination should repeat the ECG twice more, and the mean of the three results should be used as the basis for judgment;
21. History of drug abuse, drug dependence, or illicit drug use within 5 years prior to screening, or positive urine drug screening;
22. Participants who consumed excessive amounts of tea, coffee, and/or caffeinated beverages (more than 8 cups per day on average, 1 cup = 200 mL) within 3 months prior to screening;
23. Participants who smoke an average of more than 5 cigarettes per day within the 3 months prior to screening;
24. Participants who frequently consume alcohol within 3 months prior to screening (i.e., weekly alcohol intake exceeding 14 units, where 1 unit = 14 g of alcohol, equivalent to 360 mL of beer, 45 mL of spirits with alcohol content of 40%, or 150 mL of wine, corresponding to 10 bottles of beer, 500 g of Baijiu, or 3 bottles of red wine per week);
25. Planned bariatric surgery, acupuncture for weight loss, liposuction, or abdominoplasty during the study; or other planned surgery during the study (except for minor surgery that, in the opinion of the investigator, does not interfere with the study);
26. Female participants who are in the lactation period within 1 month prior to screening or during the study; or female participants with positive result in pregnancy test;
27. Participants who have engaged in unprotected sexual intercourse within 14 days prior to study treatment (applicable to female participants only);
28. Participants with history of needle phobia or blood phobia, or participants assessed by the investigator as having difficulty in blood collection, or participants cannot tolerate blood collection via venipuncture/indwelling needle;
29. Other participants deemed unsuitable for participating in the study by the investigator or participants who voluntarily withdraw from the study or who are lost to follow-up for personal reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
To evaluate the bioequivalence of HS-20094 MDV pen and AI pen following multiple doses at 15 mg. | From Day 1 to Day 169
  PK parameters of HS-20094 following multiple doses at 15 mg administered via HS-20094 MDV pen and AI pen: AUC0-168h.
To evaluate the bioequivalence of HS-20094 MDV pen and AI pen following multiple doses at 15 mg. | From Day 1 to Day 169
  PK parameters of HS-20094 following multiple doses at 15 mg administered via HS-20094 MDV pen and AI pen: Cmax

SECONDARY OUTCOMES:
To evaluate the bioequivalence of HS-20094 MDV pen and AI pen following multiple doses at 10 mg | From Day 1 to Day 169
  PK parameters following multiple doses at 10 mg administered via the HS-20094 MDV pen and AI pen: AUC0-168h;
To evaluate the bioequivalence of HS-20094 MDV pen and AI pen following multiple doses at 10 mg | From Day 1 to Day 169
  PK parameters following multiple doses at 10 mg administered via the HS-20094 MDV pen and AI pen: Cmax
To evaluate the safety following administration via the HS-20094 MDV pen and AI pen | From Day 1 to Day 204
  Adverse events
Number of participants with Vital signs | From Day 1 to Day 204
  To evaluate the safety following administration via the HS-20094 MDV pen and AI pen
To evaluate the safety following administration via the HS-20094 MDV pen and AI pen | From Day 1 to Day 204
  Number of participants with Abnormal Laboratory Values
To evaluate the safety following administration via the HS-20094 MDV pen and AI pen | From Day 1 to Day 204
  12-lead ECG, including heart rate, P-R interval, RR interval, QRS, and QTcF
To evaluate the safety following administration via the HS-20094 MDV pen and AI pen | From Day 1 to Day 204
  Physical examination questionnaire includes: general appearance, skin, lymph nodes, head, throat/thyroid, chest, abdomen, musculoskeletal system, nervous system, cardiovascular system, and others.
To evaluate the immunogenicity of HS-20094 MDV pen and AI pen after treatment. | Days 1, 29, 57, 85, 106, 141, and 169
  ADA of HS-20094: ADA positivity rate
To evaluate the immunogenicity of HS-20094 MDV pen and AI pen after treatment. | Days 1, 29, 57, 85, 106, 141, and 169
  ADA of HS-20094: Including ADA titer.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China